CLINICAL TRIAL: NCT00769002
Title: Impact of Bilateral Priming on Response to Unilateral Flu Vaccination
Brief Title: PET-CT Scans in Healthy Volunteers After Flu Vaccination
Acronym: Pro00000226
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00000226 - R21AI077102; 5R21AI077102-03 (NIH)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Flu
Keywords: influenza; flu; vaccine; vaccination; immune response; FluShield; FluMist; PET-CT; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Natural Infection (Active Comparator): previously naturally infected
  Interventions: Biological: FluShield; Procedure: Blood Draws; Procedure: FDG PET-CT Scan; Genetic: Cytokine Profiling
- FluShield - influenza positivity (Active Comparator): prior FluShield ipsilateral vaccinated
  Interventions: Biological: FluShield; Biological: FluShield - same arm; Procedure: Blood Draws; Procedure: FDG PET-CT Scan; Genetic: Cytokine Profiling
- FluShield - influenza positivity2 (Active Comparator): prior FluShield contralateral vaccinated
  Interventions: Biological: FluShield; Biological: FluShield - opposite arm; Procedure: Blood Draws; Procedure: FDG PET-CT Scan; Genetic: Cytokine Profiling
- FluMist (Active Comparator): prior FluMist vaccinated.
  Interventions: Biological: FluShield; Procedure: Blood Draws; Procedure: FDG PET-CT Scan; Genetic: Cytokine Profiling

INTERVENTIONS:
Biological: FluShield — Flu vaccine
Biological: FluShield - same arm — Flu vaccine
  Arms: FluShield - influenza positivity
Biological: FluShield - opposite arm — Flu vaccine
  Arms: FluShield - influenza positivity2
Procedure: Blood Draws — 50 cc of heparinized blood and 10 cc of serum at study entry and at 10-12 week post vaccination
Procedure: FDG PET-CT Scan — PET scan
Genetic: Cytokine Profiling — Blood draw for Cytokine Profiling Draw at 2,4 and 6 weeks post vaccination

SUMMARY:
This study is being done to learn how previous flu vaccination or previous infection with flu virus affects the immune response to vaccination.

DETAILED DESCRIPTION:
Until recently, all recipients of influenza vaccine received a killed form of virus, typically in the same nondominant arm, each year before flu season. We hypothesize that natural infection, and some forms of vaccination, could allow vaccine induced responses to spread beyond the local lymph nodes near the vaccination site. From a practical perspective, if vaccine induced proliferation of specific immune cells in sites distant from the vaccination site lead to beneficial immune memory, it would suggest vaccination strategies that could be as simple as alternating the injected arm from year to year, or alternating inhaled vs. injected forms of vaccine.

This will be a 4 armed prospective study of individuals receiving unilateral FluShield i.m. Healthy adult volunteers 21-55 will be grouped according to the following criteria: I. Documented history of prior natural infection with influenza A or B within the past 5 years (diagnostic test or high titer hemagglutinin HA Ab in absence of vaccination); II. History of FluMist vaccination within the past 2 years; III. History of TIV (Trivalent (Inactivated) Influenza Vaccine) vaccination, any number of times, but only in a single (e.g., non-dominant) arm. Within one month of screening and baseline blood draws for PBMCs (Peripheral blood mononuclear cells) and Ab (antibody) titers, individuals will receive FluShield injections. For those individuals with prior history of unilateral TIV injections, half will receive their shots in the same arm that has always been injected (Group IIIa). The other half of these individuals will receive Flushield in the opposite (dominant) arm (Group IIIb).

Upon entering the study, 50cc of heparinized blood and 10 cc of serum will be drawn by antecubital venipuncture. Within 4 weeks of this blood draw, volunteers will receive a standard dose of i.m. TIV (FluShield). Four-seven days later they will have an FDG PET-CT scan performed after an 8 hour fast.

Additional blood draws of 50cc heparinized blood and 10 cc serum will be obtained at 2, 4, and 6 weeks post vaccination, and at 10-12 months post vaccination. After the last blood draw, volunteers will also be asked questions pertaining to flu-like symptoms during the past 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 21-55 years old.
* Willingness to participate in the study for a full year including multiple blood draws and PET-CT scanning

Exclusion Criteria:

* Diabetes
* Use of systemic steroids
* Pregnancy or unwillingness to practice birth control of some kind through the PET-CT scanning period
* Recent vaccination for other reasons (e.g., traveler's vaccines)
* Significant intercurrent illness that might interfere with vaccination "take" or interpretation of PET-CT scanning (e.g., chemotherapy for cancer)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schwartz, MD, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univarsity medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PET-CT Scan Influenza Vaccine Response: Previous influenza positivity
  FluShield, FluMist: Flu vaccine
  Previous influenza positivity
  Primary Outcome Measure:
  1. Not Posted PET-CT Scan [Time Frame: 4-7 days after flu vaccine]
     Secondary Outcome Measures:
  2. Not Posted Cytokine Profiling [Time Frame: 2-6 weeks and 10-12 months post flu vaccination Active Comparator: Cytokine Profiling FluShield, FluMist No previous influenza positivity
  Primary Outcome Measure:
  1. Not Posted PET-CT Scan [Time Frame: 4-7 days after flu vaccine]
     Secondary Outcome Measures:
  2. Not Posted Cytokine Profiling [Time Frame: 2-6 weeks and 10-12 months post flu vaccination
- Cytokine Profiling: No previous influenza positivity
  FluShield, FluMist: Flu vaccine
  Primary Outcome Measure:
  1. Not Posted PET-CT Scan [Time Frame: 4-7 days after flu vaccine]
     Secondary Outcome Measures:
  2. Not Posted Cytokine Profiling [Time Frame: 2-6 weeks and 10-12 months post flu vaccination Active Comparator: Cytokine Profiling FluShield, FluMist No previous influenza positivity
  Primary Outcome Measure:
  1. Not Posted PET-CT Scan [Time Frame: 4-7 days after flu vaccine]
     Secondary Outcome Measures:
  2. Not Posted Cytokine Profiling [Time Frame: 2-6 weeks and 10-12 months post flu vaccination
Period: Overall Study
Arm/Group | PET-CT Scan Influenza Vaccine Response | Cytokine Profiling
Started | 9 | 9
Completed | 0 | 0
Not Completed | 9 | 9
Not completed — Study was not completed, no data | 9 | 9

BASELINE CHARACTERISTICS:
Population: This study was not completed as planned, and data collected is not available despite all efforts as the PI has left the institution. Additionally, no manuscript, or study report was developed and therefore no data available to confirm the validity of or address the comments in relation to the previously entered results information.
Groups:
- Influenza Vaccine FluShield, FluMist: Group I - Previous influenza positivity A or B within the past 5 years
- Cytokine Profiling FluShield, FluMist: Group II - History of FluMist vaccination within the past 2 years
- Unilateral TIV Injections FluShield: Group III a - History of TIV vaccination, any number of times, but only in a single (e.g., non-dominant) arm. For those individuals with prior history of unilateral TIV injections, half will receive their shots in the same arm that has always been injected (Group IIIa).
- Opposite Arm FluShield: Group IIIb - Within one month of screening and baseline blood draws for PBMCs and Ab titers, individuals will receive FluShield injections. The other half of these individuals will receive Flushield in the opposite (dominant) arm (Group IIIb).
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine FluShield, FluMist | Cytokine Profiling FluShield, FluMist | Unilateral TIV Injections FluShield | Opposite Arm FluShield | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Categorical — Men and women ages 21-55
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: PET Scan AB Response
Description: Natural infection but not ipsilateral IM injection of FluShield, will prime the host for a specific activation of spleen and bilateral lymph nodes following a subsequent i.m injection of FluShield, as detected by PET-CT performed 4-7 days post- FluShield immunization.
Time Frame: 4-7 days
Population: as for baseline characteristics
Arm/Group | PET-CT Scan Influenza Vaccine Response
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Influenza Vaccine FluShield, FluMist: Previous influenza positivity
  Primary Outcome Measure:
  1. PET-CT Scan [Time Frame: 4-7 days after flu vaccine]
     Secondary Outcome Measures:
  2. Cytokine Profiling [Time Frame: 2-6 weeks and 10-12 months post flu vaccination
  FluShield, FluMist: Flu vaccine
- Cytokine Profiling FluShield, FluMist: No previous influenza positivity
  Primary Outcome Measure:
  1. PET-CT Scan [Time Frame: 4-7 days after flu vaccine]
     Secondary Outcome Measures:
  2. Cytokine Profiling [Time Frame: 2-6 weeks and 10-12 months post flu vaccination
  FluShield, FluMist: Flu vaccine
Arm/Group | Influenza Vaccine FluShield, FluMist | Cytokine Profiling FluShield, FluMist
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
This study was not completed and data collected is not available despite all efforts as PI has left the institution. No manuscript/study report was developed and there are no data to confirm validity or address comments in previously entered results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes